CLINICAL TRIAL: NCT03359200
Title: Analysis of the Microbiota in Goldmann Applanation Tonometers at a Reference Service in Goiânia
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: Tonometro ARVO
Record Dates: First submitted 2017-11-25; First posted 2017-12-02 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the microbiota of goldmann tonometers and its possible change over the visits

ELIGIBILITY:
Inclusion Criteria:

* collection of material in the period

Exclusion Criteria:

* collection of material out of the period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: no patient was studied
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Analysis of the microbiota in tonometers performed by means of swab collections | 1 month
  collect swabs of the tonometers before and after the visits to evaluate the change of the microbiota and, therefore, to evaluate the effectiveness of the asepsis.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No